CLINICAL TRIAL: NCT07267416
Title: Prospective Randomized Controlled Study on the Impact of Combined PSi + NIRS Monitoring in the Prevention of Postoperative Cognitive Disorders in Cardiac Surgery.
Brief Title: Impact of Combined PSi + NIRS Monitoring in the Prevention of Postoperative Cognitive Disorders in Cardiac Surgery.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Tatiana Besse-Hammer, Head of Clinical Research Unit, Brugmann University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PsiNIRS
Record Dates: First submitted 2025-11-25; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Cognitive Disorders
MeSH Terms: conditions — Postoperative Cognitive Complications | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard monitoring + NIRS (Experimental): Dual intraoperative cerebral monitoring, consisting of
  * PSi (Patient State Index) via SedLine®, an indicator of anesthetic depth (normal values between 25 and 50),
  * NIRS (Near Infrared Spectroscopy), real-time measurement of regional cerebral oxygenation, associated with a standardized therapeutic algorithm.
  Interventions: Device: NIRS (Near Infrared Spectroscopy); Device: SedLine®
- Standard monitoring (Active Comparator): Intraoperative cerebral monitoring, consisting of PSi (Patient State Index) via SedLine®.
  Interventions: Device: SedLine®

INTERVENTIONS:
Device: NIRS (Near Infrared Spectroscopy) — Real-time measurement of regional cerebral oxygenation.
  Arms: Standard monitoring + NIRS
Device: SedLine® — The SedLine® Brain Function Monitoring device (Masimo Corporation, model RDS7A, CE certified) uses four forehead electrodes to record EEG activity. The Patient State Index (PSi), calculated in real time, is interpreted within a target range of 25 to 50 to ensure adequate general anesthesia. The device complies with international standards for electrical safety (IEC 60601) and hospital use.

SUMMARY:
Advances in cardiac medicine and anesthesia have made it possible to expand the indications for open heart surgery to increasingly older and more complex patients. This development is taking place in a demographic context where the aging of the world population has become a structural reality. However, postoperative neurocognitive complications, and in particular postoperative cognitive disorders (POCD), are not limited to the elderly. They can affect all adults, including younger adults, particularly in the presence of risk factors such as prolonged cardiopulmonary bypass, deep anesthesia, or episodes of intraoperative cerebral desaturation.

The PSi-NIRS study was designed with this broad perspective in mind. It will include all adult patients (≥18 years) eligible for cardiac surgery under extracorporeal circulation, with a secondary analysis dedicated to patients aged 65 years and older, a group in which POCD is more frequent, more long-lasting, and often has more serious consequences. This division will allow to assess the impact of cerebral monitoring both in the general adult population and within a well-defined geriatric subgroup.

The pathophysiological mechanisms involved in POCD are now better understood. On the one hand, insufficient cerebral oxygenation, even transient, can disrupt neuronal homeostasis for a prolonged period. On the other hand, excessively deep anesthesia, leading to periods of EEG suppression, is recognized as a risk marker for delirium and postoperative cognitive decline. These two dimensions - perfusion and cortical activity - constitute complementary targets for prevention.

Independently of each other, two tools available today - near-infrared spectroscopy (NIRS) and processed electroencephalography (PSi via SedLine®) - have shown their value in cardiac surgery. The use of NIRS to guide intraoperative adjustments has been associated with a reduction in neurological complications. Anesthetic guidance by EEG makes it possible to limit periods of suppression, linked to an increased risk of delirium and POCD. However, to date, no randomized study has evaluated the combined and coordinated use of these two modalities, with a predefined therapeutic algorithm allowing real-time clinical intervention based on critical thresholds.

The PSi-NIRS study is therefore part of a logic of scientific continuity, but takes a methodological step forward by testing for the first time an integrated and proactive approach to cerebral monitoring, applied to a surgical context with high neurological risk. It aims to verify whether this strategy can improve the postoperative cognitive trajectory of patients, in the short and medium term, by targeting the real points of intraoperative cerebral vulnerability.

ELIGIBILITY:
Inclusion Criteria:

* Elective or relatively emergency surgery for valve surgery (pulmonary or tricuspid valves) or coronary artery bypass grafting (CABG)
* Preoperative cognitive assessment MoCA ≥ 20 (during the preoperative consultation if applicable or on day 1)
* ASA score II to IV

Exclusion Criteria:

* History of sequelae of stroke
* Diagnosis or strong suspicion of dementia (according to DSM-V criteria).
* Preoperative encephalopathy
* Severe chronic renal failure requiring dialysis
* Patients with chronic respiratory failure who are oxygen-dependent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
MoCA (Montreal Cognitive Assessment) | Baseline, pre-surgery
  Rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation.The total possible score is 30 points; a score of 26 or above is considered normal.
MoCA (Montreal Cognitive Assessment) | 2 days post surgery
  Rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation.The total possible score is 30 points; a score of 26 or above is considered normal.
MoCA (Montreal Cognitive Assessment) | 7 days post surgery
  Rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation.The total possible score is 30 points; a score of 26 or above is considered normal.
MoCA (Montreal Cognitive Assessment) | 25 days post surgery
  Rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation.The total possible score is 30 points; a score of 26 or above is considered normal.
MoCA (Montreal Cognitive Assessment) | 30 days post surgery
  Rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation.The total possible score is 30 points; a score of 26 or above is considered normal.

SECONDARY OUTCOMES:
Postoperative length of stay | Immediately after the surgery
  Postoperative length of stay
Cumulative duration of burst deletions (SedLine) | During the surgery
Cumulative duration of NIRS desaturation episodes | During the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Aimane MENIOUI, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No